CLINICAL TRIAL: NCT03132883
Title: Evolution of Indications for Transbronchial Ganglionic Ultrasound in the Picardie Region Over the Period 2008 - 2013
Brief Title: Evolution of Indications for Transbronchial Ganglionic Ultrasound
Acronym: EBUSPicardie
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-41 Dr Basille-2
Record Dates: First submitted 2017-04-14; First posted 2017-04-28 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Transbronchial Surgery; Lymph Node Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
New indications for bronchial echo-endoscopies with transbronchial needle aspiration (EBUS-PTBA) have appeared since the first French centers with this technique were fitted. Evaluate the respective share of each indication of EBUS-AWPB over time over the period 2008 - 2013

DETAILED DESCRIPTION:
Transbronchial puncture is a technique known for many years with the first description found in 1949 by Shieppati. Subsequently, this technique allowing an exploration of the mediastinal lymph nodes became widespread with the work of Wang in 1983. However, the need to have exact knowledge of the different puncture sites in order to obtain maximum profitability with this examination in particular In staging and diagnosis in bronchopulmonary cancers (CBP) explains a significant difference in profitability between operators based on their experience. It was not until 1990 that Germans coupled the technique of radial ultrasound with that of bronchoscopy by introducing a balloon catheter inflated with a liquid allowing the best transmission of ultrasound. It is the German team of Herth who developed this technique in 1999 under the name of bronchial echo-endoscopy (EBUS). The association of echo-endoscopy before transbronchial punctures significantly improves the performance of the examination. In 2004, Yasufusu shows the interest of the real-time visualization of the lymph nodes for the marking as well as the punctures. Therefore, the indications for bronchial echoendoscopies with transbronchial needle puncture (EBUS-PTBA) are precisely defined in the nodal staging of CBP with good profitability and a reduction in surgical mediastinoscopy. Then, over time, there is an extension of indications with the diagnosis of Non-Small Cell Lung Broncho-Pulmonary Cancers (NSCLC) or Small Cell Broncho-Pulmonary Cancers (CBPC), the diagnosis of ganglion metastases of extra-thoracic primary tumors , Diagnosis of sarcoidosis or other more anecdotal uses (tuberculosis, lymphoma).

Two Picard centers were among the first in France to be equipped with echoendoscopes (2007 for the CH of Saint Quentin and 2008 for the CHU of Amiens). This allows our two centers to have a fairly consistent retreat on the technique since its implantation in France. While many studies are concerned with one or other indication in isolation, there is no study to the best of our knowledge relating the evolution over time of the respective share of each of these indications in daily practice . Given the current multiplication of potential indications for EBUS-PTBA, it seems interesting to analyze the place of these new indications in the daily activity of endoscopic centers equipped with an echo-endoscope. The main objective is to evaluate the respective share of each indication over time over the study period. Secondary objectives are the evaluation of the diagnostic performance of EBUS-PTBA, the evaluation of the abusively carried-out EBUS-PTBA (examination carried out for purely diagnostic purposes, whereas conventional bronchial fibroscopy Diagnosis of certainty) and evaluation of concordance between EBUS-PTBA and surgery in CBP staging indications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a first linear echo-endoscopy at the CHU of Amiens and the CH of Saint-Quentin between January 2008 and December 2013

Exclusion Criteria:

* Patient sent by a center outside Picardie
* Patient having expressed a refusal to participate in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusive patients will be made from the computer database of endoscopy services of each of the 2 centers listing endoscopic examinations carried out over the period of interest
Sampling Method: Non-Probability Sample
Enrollment: 1036 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Analysis of endoscopic examination (EBUS-PTBA): analysis of diagnosis and / or staging of bronchial carcinoma, diagnosis of sarcoidosis, tuberculosis, lymphoma, staging of extra-thoracic tumors | 5 years
  Analysis of endoscopic examination (EBUS-PTBA): analysis of diagnosis and / or staging of bronchial carcinoma, diagnosis of sarcoidosis, tuberculosis, lymphoma, staging of extra-thoracic tumors

CONTACTS AND LOCATIONS:
Overall Officials: Damien BASILLE, Dr, Principal Investigator — CHU AMIENS PICARDIE
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France